CLINICAL TRIAL: NCT01946204
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Study of ARN-509 in Men With Non-Metastatic (M0) Castration-Resistant Prostate Cancer
Brief Title: A Study of Apalutamide (ARN-509) in Men With Non-Metastatic Castration-Resistant Prostate Cancer
Acronym: SPARTAN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR102931; ARN-509-003; 56021927PCR1007 (Other: Janssen Research & Development, LLC); 2012-004322-24 (EudraCT Number)
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate neoplasms; Prostate cancer; Castration-resistant prostate cancer; Non-metastatic castration-resistant prostate cancer; ARN-509; Apalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A: Apalutamide (Experimental)
  Interventions: Drug: Apalutamide
- Treatment Arm B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apalutamide — 240 mg tablets administered by mouth on a continuous once daily dosing regimen
  Arms: Treatment Arm A: Apalutamide
Drug: Placebo — Matched placebo tablets administered by mouth on a continuous once daily dosing regimen
  Arms: Treatment Arm B: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of apalutamide in adult men with high-risk non-metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This Phase 3 clinical trial is an essential step in the evaluation of an investigational medication to see if it may be useful in treating prostate cancer. The purpose of the SPARTAN study is to compare the safety and effectiveness of the investigational medication to placebo in delaying prostate cancer from spreading to other parts of the body. A placebo is a pill that looks like the investigational medication but does not contain any active medication, a dummy pill.

Phase 3 studies are performed after preliminary evidence suggesting effectiveness of the drug has been obtained in previous Phase 2 studies. These studies are intended to gather the additional information about effectiveness and safety that is needed to evaluate the overall benefit-risk relationship of the drug.

Study participants will take the oral investigational medication daily. One cycle of study treatment lasts 4 weeks or 28 days. The number of cycles will depend on how you and your cancer respond to the study medication.

In order for the researchers to evaluate and compare the study results, there are two different study groups. Study participants will be randomly (like flipping a coin) assigned to one of these groups:

* One group will receive their current treatment along with the investigational medication
* One group will receive their current medications along with a placebo

The investigational medication will be given to 2 out of every 3 study participants. Neither you nor the study staff will know which group you are in. However, in case of a medical emergency, your study doctor can quickly find out which treatment group you are in.

All participants will continue to receive their current treatment along with either the investigational medication or a placebo. The selections will be random, and you may remain on investigational treatment until your disease worsens, or until significant side effects occur or you can no longer tolerate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features with high risk for development of metastases, defined as prostate-specific antigen doubling time (PSADT) less than or equal to (<=) 10 months. PSADT is calculated using at least 3 prostate-specific antigen (PSA) values obtained during continuous ADT (androgen deprivation therapy)
* Castration-resistant prostate cancer demonstrated during continuous ADT, defined as 3 PSA rises, at least 1 week apart, with the last PSA greater than (>) 2 nanogram per milliliter (ng/mL)
* Maintain castrate levels of testosterone within 4 weeks prior to randomization and throughout the study
* Patients currently receiving bone loss prevention treatment with bone-sparing agents must be on stable doses for at least 4 weeks prior to randomization
* Patients who received a first generation anti-androgen (for example, bicalutamide, flutamide, nilutamide) must have at least a 4-week washout prior to randomization AND must show continuing disease (PSA) progression (an increase in PSA) after washout
* At least 4 weeks must have elapsed from the use of 5-alpha reductase inhibitors, estrogens, and any other anti-cancer therapy prior to randomization
* At least 4 weeks must have elapsed from major surgery or radiation therapy prior to randomization
* Eastern Cooperative Oncology Group Performance Status 0 or 1
* Resolution of all acute toxic effects of prior therapy or surgical procedure to Grade <= 1 or baseline prior to randomization
* Adequate organ function according to protocol-defined criteria
* Administration of growth factors or blood transfusions will not be allowed within 4 weeks of the hematology labs required to confirm eligibility

Exclusion Criteria:

* Presence of confirmed distant metastases, including central nervous system and vertebral or meningeal involvement
* Symptomatic local or regional disease requiring medical intervention
* Prior treatment with second generation anti-androgens
* Prior treatment with CYP17 inhibitors
* Prior treatment with radiopharmaceutical agents, or any other investigational agent for non-metastatic castration-resistant prostate cancer
* Prior chemotherapy for prostate cancer except if administered in the adjuvant/neoadjuvant setting
* History of seizure or condition that may pre-dispose to seizure
* Concurrent therapy with protocol-defined excluded medications
* History or evidence of any of the following conditions: any prior malignancy (other than adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) within 5 years prior to randomization; severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events, or clinically significant ventricular arrhythmias within 6 months prior to randomization; uncontrolled hypertension; gastrointestinal disorder affecting absorption; active infection; and, any other condition that, in the opinion of the investigator, would impair the patient's ability to comply with study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1207 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aragon Pharmaceuticals, Inc. Clinical Trial, Study Director — Aragon Pharmaceuticals, Inc.
Locations (379):
- United States (122):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Chandler, Arizona
  - Tucson, Arizona
  - Duarte, California
  - Fullerton, California
  - Laguna Woods, California
  - Los Angeles, California
  - Orange, California
  - Roseville, California
  - Sacramento, California
  - San Bernardino, California
  - San Diego, California
  - San Francisco, California
  - Santa Monica, California
  - Sherman Oaks, California
  - Stanford, California
  - Tarzana, California
  - Torrance, California
  - Denver, Colorado
  - Englewood, Colorado
  - Glenwood Springs, Colorado
  - Grand Junction, Colorado
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Boca Raton, Florida
  - Bradenton, Florida
  - Daytona Beach, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Wellington, Florida
  - Meridian, Idaho
  - Chicago, Illinois
  - Decatur, Illinois
  - Maywood, Illinois
  - Melrose Park, Illinois
  - Carmel, Indiana
  - Jeffersonville, Indiana
  - Muncie, Indiana
  - West Des Moines, Iowa
  - Westwood, Kansas
  - Wichita, Kansas
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Rockville, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Lansing, Michigan
  - Minneapolis, Michigan
  - Royal Oak, Michigan
  - Duluth, Minnesota
  - Bay Saint Louis, Mississippi
  - Southaven, Mississippi
  - Kansas City, Missouri
  - Missoula, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Hooksett, New Hampshire
  - Hackensack, New Jersey
  - Lawrenceville, New Jersey
  - Morristown, New Jersey
  - Mount Laurel, New Jersey
  - New Brunswick, New Jersey
  - Voorhees Township, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Mineola, New York
  - New York, New York
  - Oneida, New York
  - Poughkeepsie, New York
  - Syracuse, New York
  - The Bronx, New York
  - Concord, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Middleburg Heights, Ohio
  - Middletown, Ohio
  - Bend, Oregon
  - Portland, Oregon
  - Tualatin, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Bryn Mawr, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - West Columbia, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Abilene, Texas
  - Amarillo, Texas
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Burien, Washington
  - Edmonds, Washington
  - Seattle, Washington
  - Tacoma, Washington
  - Green Bay, Wisconsin
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (17):
  - Adelaide
  - Box Hill
  - Camperdown
  - Darlinghurst
  - Geelong
  - Gosford
  - Hobart
  - Kogarah
  - Liverpool
  - Melbourne
  - Nedlands
  - Parkville
  - South Woodville
  - Southport
  - Sydney
  - Tweed Heads
  - Wollongong
- Austria (4):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Belgium (6):
  - Brussels
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
  - Ottignies
- Canada (27):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Abbotsford, British Columbia
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Moncton, New Brunswick
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Brampton, Ontario
  - Brantford, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - North York, Ontario
  - Oakville, Ontario
  - Ottawa, Ontario
  - Owen Sound, Ontario
  - Toronto, Ontario
  - Gatineau, Quebec
  - Granby, Quebec
  - Greenfield Park, Quebec
  - Laval, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- Czechia (5):
  - Liberec
  - Olomouc
  - Opava
  - Pilsen
  - Prague
- Denmark (4):
  - Aalborg C
  - Copenhagen
  - Odense
  - Roskilde
- Finland (5):
  - Helsinki
  - Oulu
  - Seinäjoki
  - Tampere
  - Turku
- France (23):
  - Angers
  - Besançon
  - Bordeaux
  - Caen Cédex 05
  - Clermont-Ferrand
  - Hyers
  - La Roche-sur-Yon
  - Le Mans
  - Lille Cedex N/a
  - Lyon
  - Marseille
  - Nice
  - Nîmes
  - Paris
  - Reims
  - Rennes
  - Rouen
  - Saint-Grégoire
  - Saint-Herblain
  - Strasbourg
  - Suresnes
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (33):
  - Aachen
  - Bergisch Gladbach
  - Berlin
  - Braunschweig
  - Cologne
  - Duisburg
  - Emmendingen
  - Frankfurt am Main
  - Göttingen
  - Greifswald
  - Hamburg
  - Hanover
  - Heidelberg
  - Heinsberg
  - Homburg/Saar
  - Jena
  - Kiel
  - Kirchheim unter Teck
  - Magdeburg
  - Mainz
  - Mannheim
  - Marburg
  - Mettmann
  - Müllheim
  - Münster
  - Nürtingen
  - Regensburg
  - Rostock
  - Tübingen
  - Weiden
  - Wilhelmshaven
  - Wuppertan
  - Zirndorf
- Hungary (5):
  - Budapest
  - Miskolc
  - Nyíregyhá
  - Sopron
  - Szentes
- Israel (7):
  - Haifa
  - Jeruselem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
  - Ẕerifin
- Japan (29):
  - Akita
  - Fukuoka
  - Gifu
  - Hakodate
  - Hiroshima
  - Hokkaido
  - Kanazawa
  - Kashiwa
  - Kita-Gun
  - Kobe
  - Koshigaya
  - Kumamoto
  - Kurume
  - Matsuyama
  - Nagano
  - Nagasaki
  - Nagoya
  - Niigata
  - Osaka
  - Ōsaka-sayama
  - Sagamihara
  - Sakura
  - Sapporo
  - Shinjuku-Ku
  - Tokushima
  - Tokyo
  - Ube
  - Wakayama
  - Yokohama
- Netherlands (6):
  - Alkmaar
  - Eindhoven
  - Hoofddorp
  - Leidschendam
  - Nijmegen
  - Rotterdam
- New Zealand (6):
  - Auckland
  - Christchurch
  - Hamilton
  - Nelson
  - Tauranga
  - Whangarei
- Nordbyhagen, Norway
- Poland (10):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Kutno
  - Lodz
  - Poznan
  - Szczecin
  - Torun
  - Warsaw
  - Wroclaw
- Romania (5):
  - Baia Mare
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Târgu Mureş
- Russia (10):
  - Barnaul
  - Ivanovo
  - Moscow
  - Obninsk
  - Omsk
  - Ryazan
  - Saint Petersburg
  - Ufa
  - Yaroslavl
  - Yekaterinburg
- Slovakia (5):
  - Banská Bystrica
  - Bratislava
  - Martin
  - Nitra
  - Trenčín
- South Korea (5):
  - Daegu
  - Gwangju
  - Pusan
  - Seongnam
  - Seoul
- Spain (19):
  - A Coruña
  - Badalona
  - Barcelona
  - Castellon
  - Girona
  - Guadalajara
  - Jerez de la Frontera
  - Las Palmas de Gran Canaria
  - Madrid
  - Málaga
  - Murcia
  - Palma de Mallorca
  - Pamplona
  - Sabadell
  - Salamanca
  - San Sebastián de los Reyes
  - Santander
  - Seville
  - Valencia
- Sweden (5):
  - Gothenburg
  - Örebro
  - Stockholm
  - Umeå
  - Uppsala
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan
- United Kingdom (16):
  - Blackburn
  - Cambridge
  - Cardiff
  - Dundee
  - Glasgow
  - Guildford
  - Leeds
  - London
  - Maidstone
  - Metropolitan Borough of Wirral
  - Nottingham
  - Plymouth
  - Southampton
  - Surrey
  - Swansea
  - Wolverhampton

REFERENCES:
- [Derived] Ni X, Sui J, Wang B, Wang H, Freedland SJ, Ye D, Zhu Y. Lower Testosterone Level and Metastases-Free Survival in Patients With Nonmetastatic Castration-Resistant Prostate Cancer Treated With Novel Antiandrogens: A Post Hoc Analysis of SPARTAN and ARAMIS. J Urol. 2025 Jul;214(1):10-17. doi: 10.1097/JU.0000000000004545. Epub 2025 Mar 25. PMID 40132221
- [Derived] Feng FY, Smith MR, Saad F, Mobadersany P, Tian SK, Yip SSF, Greshock J, Khan N, Yu MK, McCarthy S, Brookman-May SD, Bourla AB, Todorovic T, Yamashita R, Huang HC, Royce TJ, Showalter TN, Griffin J, Mitani A, Esteva A, Small EJ. Digital Pathology-Based Multimodal Artificial Intelligence Scores and Outcomes in a Randomized Phase III Trial in Men With Nonmetastatic Castration-Resistant Prostate Cancer. JCO Precis Oncol. 2025 Jan;9:e2400653. doi: 10.1200/PO-24-00653. Epub 2025 Jan 31. PMID 39889245
- [Derived] Roy S, Malone S, Wing K, Chowdhury S, Kishan AU, Sun Y, Wallis CJD, Mohamad O, Jia AY, Swami U, Zaorsky NG, Morgan SC, Ong M, Agarwal N, Spratt DE, Small EJ, Saad F. Prior Local Therapy and First-Line Apalutamide in Patients With Nonmetastatic Castration-Resistant Prostate Cancer: A Secondary Analysis of the SPARTAN Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2439434. doi: 10.1001/jamanetworkopen.2024.39434. PMID 39405060
- [Derived] Karsh LI, Bevans KB, Saad F, Chung BH, Oudard S, Brookman-May SD, McCarthy SA, Smith MR, Chi KN, Small EJ, Agarwal N. Prostate-specific antigen and health-related quality of life in individuals with advanced prostate cancer treated with apalutamide: a plain language summary of the SPARTAN and TITAN studies. Future Oncol. 2024;20(35):2689-2698. doi: 10.1080/14796694.2024.2384257. Epub 2024 Aug 20. PMID 39163505
- [Derived] Shen J, Chowdhury S, Agarwal N, Karsh LI, Oudard S, Gartrell BA, Feyerabend S, Saad F, Pieczonka CM, Chi KN, Brookman-May SD, Rooney B, Bhaumik A, McCarthy SA, Bevans KB, Mundle SD, Small EJ, Smith MR, Graff JN. Apalutamide efficacy, safety and wellbeing in older patients with advanced prostate cancer from Phase 3 randomised clinical studies TITAN and SPARTAN. Br J Cancer. 2024 Jan;130(1):73-81. doi: 10.1038/s41416-023-02492-8. Epub 2023 Nov 11. PMID 37951974
- [Derived] Pollock Y, Smith MR, Saad F, Chowdhury S, Oudard S, Hadaschik B, Olmos D, Lee JY, Uemura H, Bhaumik A, Londhe A, Rooney B, Brookman-May SD, De Porre P, Mundle SD, Small EJ. Clinical characteristics associated with falls in patients with non-metastatic castration-resistant prostate cancer treated with apalutamide. Prostate Cancer Prostatic Dis. 2023 Mar;26(1):156-161. doi: 10.1038/s41391-022-00592-9. Epub 2022 Oct 8. PMID 36209239
- [Derived] Chowdhury S, Oudard S, Uemura H, Joniau S, Dearden L, Capone C, Van Sanden S, Diels J, Hadaschik BA. Apalutamide Compared with Darolutamide for the Treatment of Non-metastatic Castration-Resistant Prostate Cancer: Efficacy and Tolerability in a Matching-Adjusted Indirect Comparison. Adv Ther. 2022 Jan;39(1):518-531. doi: 10.1007/s12325-021-01885-6. Epub 2021 Nov 19. PMID 34797506
- [Derived] Uemura H, Koroki Y, Iwaki Y, Imanaka K, Kambara T, Lopez-Gitlitz A, Smith A, Uemura H. Skin rash following Administration of Apalutamide in Japanese patients with Advanced Prostate Cancer: an integrated analysis of the phase 3 SPARTAN and TITAN studies and a phase 1 open-label study. BMC Urol. 2020 Sep 2;20(1):139. doi: 10.1186/s12894-020-00689-0. PMID 32878613
- [Derived] Smith MR, Mehra M, Nair S, Lawson J, Small EJ. Relationship Between Metastasis-free Survival and Overall Survival in Patients With Nonmetastatic Castration-resistant Prostate Cancer. Clin Genitourin Cancer. 2020 Apr;18(2):e180-e189. doi: 10.1016/j.clgc.2019.10.030. Epub 2019 Nov 6. PMID 31980408
- [Derived] Saad F, Cella D, Basch E, Hadaschik BA, Mainwaring PN, Oudard S, Graff JN, McQuarrie K, Li S, Hudgens S, Lawson J, Lopez-Gitlitz A, Yu MK, Smith MR, Small EJ. Effect of apalutamide on health-related quality of life in patients with non-metastatic castration-resistant prostate cancer: an analysis of the SPARTAN randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2018 Oct;19(10):1404-1416. doi: 10.1016/S1470-2045(18)30456-X. Epub 2018 Sep 10. PMID 30213449
- [Derived] Smith MR, Saad F, Chowdhury S, Oudard S, Hadaschik BA, Graff JN, Olmos D, Mainwaring PN, Lee JY, Uemura H, Lopez-Gitlitz A, Trudel GC, Espina BM, Shu Y, Park YC, Rackoff WR, Yu MK, Small EJ; SPARTAN Investigators. Apalutamide Treatment and Metastasis-free Survival in Prostate Cancer. N Engl J Med. 2018 Apr 12;378(15):1408-1418. doi: 10.1056/NEJMoa1715546. Epub 2018 Feb 8. PMID 29420164

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received apalutamide matched placebo tablets orally on a continuous once daily dosing regimen along with androgen deprivation therapy (ADT) until disease progression, withdrawal of consent or unacceptable toxicity or death.
- Apalutamide: Participants received apalutamide orally at a starting dose of 240 milligram (mg) (8 x 30 mg capsules then 4 x 60 mg tablets) in a continuous treatment cycles (each treatment cycle is of 28 days) once daily dosing regimen along with androgen deprivation therapy (ADT) until disease progression, withdrawal of consent or unacceptable toxicity or death.
Period: Overall Study
Arm/Group | Placebo | Apalutamide
Started | 401 | 806
Treated | 398 | 803
Completed | 0 | 0
Not Completed | 401 | 806
Not completed — Death | 38 | 59
Not completed — Withdrawal by Subject | 37 | 50
Not completed — Lost to Follow-up | 3 | 7
Not completed — Ongoing | 316 | 687
Not completed — Other | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Apalutamide | Total
Number analyzed (Participants) | 401 | 806 | 1207
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (7.92) | 73.7 (8.07) | 73.9 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 401 | 806 | 1207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 11 | 16
  Not Hispanic or Latino | 338 | 659 | 997
  Unknown or Not Reported | 58 | 136 | 194
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 47 | 93 | 140
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 48 | 68
  White | 276 | 524 | 800
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 58 | 136 | 194
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 11 | 30 | 41
  Austria | 2 | 4 | 6
  Belgium | 3 | 4 | 7
  Canada | 21 | 61 | 82
  Czech Republic | 14 | 20 | 34
  Denmark | 7 | 14 | 21
  Finland | 5 | 7 | 12
  France | 21 | 39 | 60
  Germany | 20 | 31 | 51
  Hungary | 1 | 4 | 5
  Israel | 7 | 7 | 14
  Italy | 12 | 24 | 36
  Japan | 21 | 34 | 55
  Netherlands | 11 | 8 | 19
  New Zealand | 2 | 6 | 8
  Norway | 3 | 4 | 7
  Poland | 6 | 28 | 34
  Romania | 5 | 7 | 12
  Russia | 11 | 24 | 35
  Slovakia | 6 | 11 | 17
  South Africa | 17 | 35 | 52
  Spain | 36 | 95 | 131
  Sweden | 3 | 10 | 13
  Taiwan, Province Of China | 5 | 14 | 19
  United Kingdom | 38 | 61 | 99
  United States | 113 | 224 | 337

OUTCOME MEASURES:

1. Secondary Outcome: Time to Metastasis (TTM)
Description: Time to metastasis (TTM) was defined as the time from randomization to the time of the scan that showed first evidence of BICR-confirmed radiographically detected bone or soft tissue distant metastasis. The TTM data for participants without metastasis were performed for US or ex-US regulatory purposes. Radiographic scans (bone scans and CT or MRI of the chest, abdomen, and pelvis) were performed for detection of metastasis throughout the study.
Time Frame: Up to approximately 43 Months
Population: ITT population included all participants who were randomized into the study, with study drug assignments designated according to initial randomization, regardless of whether participants received what was assigned.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Apalutamide
Number analyzed (Participants) | 401 | 806
Months
  US Regulatory | 16.59 [14.59 to 18.46] | 40.51 [NA to NA] — NA signifies: lower and upper limit of CI was not estimable (NA) as lower, or upper, or both limits of CI for survivor function were above 0.5 using log(-log) transformation (default of SAS Proc Lifetest).
  EX-US Regulatory | 15.70 [14.55 to 18.40] | 40.51 [31.15 to 40.51]
Statistical Analysis 1: Comparison: Placebo vs Apalutamide; Statistical Analysis for TTM by BICR (US Regulatory); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.271, 95% CI 2-sided [0.219 to 0.335]
Statistical Analysis 2: Comparison: Placebo vs Apalutamide; Statistical Analysis for TTM by BICR (Ex-US Regulatory); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.279, 95% CI 2-sided [0.227 to 0.342]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS defined as time from randomization to first documentation of BICR-confirmed radiographic progressive disease (PD) (development of distant/local/regional metastasis)/death due to any cause whichever occurred first. PFS data for participants without loco-regional disease were performed for US/ex-US regulatory purposes. Radiographic scans (bone scans and CT/MRI of chest,abdomen,pelvis) performed for detection of metastasis throughout study. PD based on RECIST v1.1; Subjects with one measurable lesion, At least 20% increase in sum of diameters of target lesions taking as reference smallest sum on study. In addition, sum must demonstrate an absolute increase of at least 5 millimeter(mm). Also, appearance of one/more new lesions was also considered PD. Subjects with non-measurable disease as per CT/MRI scans, unequivocal progression/appearance of one or more new lesions was considered PD. For new bone lesions detected on bone scans, second imaging (CT/MRI) was required to confirm PD.
Time Frame: Up to approximately 43 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Apalutamide
Number analyzed (Participants) | 401 | 806
Months
  US Regulatory | 14.72 [14.49 to 18.37] | 40.51 [NA to NA] — NA signifies: lower and upper limit of CI was not estimable (NA) as lower, or upper, or both limits of CI for survivor function were above 0.5 using log(-log) transformation (default of SAS Proc Lifetest).
  EX-US Regulatory | 14.65 [11.27 to 17.97] | 40.51 [29.40 to 40.51]
Statistical Analysis 1: Comparison: Placebo vs Apalutamide; Statistical Analysis for PFS by BICR (US Regulatory); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.291, 95% CI 2-sided [0.238 to 0.356]
Statistical Analysis 2: Comparison: Placebo vs Apalutamide; Statistical Analysis for PFS by BICR (EX-US Regulatory); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.300, 95% CI 2-sided [0.247 to 0.364]

3. Secondary Outcome: Time to Symptomatic Progression
Description: Time to symptomatic progression was defined as the time from randomization to documentation in the CRF of any of the following (whichever occurred earlier): a) development of a skeletal-related event (pathologic fracture, spinal cord compression, or need for surgical intervention or radiation therapy to the bone); b) pain progression or worsening of disease-related symptoms requiring initiation of a new systemic anti-cancer therapy; or c) development of clinically significant symptoms due to loco-regional tumor progression requiring surgical intervention or radiation therapy.
Time Frame: Up to approximately 43 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Apalutamide
Number analyzed (Participants) | 401 | 806
Months | NA [36.83 to NA] — NA signifies: median and upper limit of CI were NA. Median was NA as KM curve did not drop to 0.5 or below. Upper limit was NA as upper limit of CI for survivor function was above 0.5 using log(-log) transformation (default of SAS Proc Lifetest). | NA [NA to NA] — The median was not estimable(NA) as Kaplan-Meier(KM) curve did not drop to 0.5 or below. The lower or upper limit was NA as lower or upper limit of CI for survivor function was above 0.5 using log(-log) transformation (default of SAS Proc Lifetest).
Statistical Analysis 1: Comparison: Placebo vs Apalutamide; Statistical Analysis for Time to Symptomatic Progression; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.447, 95% CI 2-sided [0.315 to 0.634]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to the date of death due to any cause.
Time Frame: Up to approximately 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Apalutamide
Number analyzed (Participants) | 401 | 806
Months | 39.03 [39.03 to NA] — Here NA signifies that the upper limit of Confidence Interval (CI) was not estimable as upper limit of CI for the survivor function was above 0.5 using log(-log) transformation (the default of SAS Proc Lifetest). | NA [NA to NA] — The median was not estimable(NA) as Kaplan-Meier(KM) curve did not drop to 0.5 or below. The lower or upper limit was NA as lower or upper limit of CI for survivor function was above 0.5 using log(-log) transformation (default of SAS Proc Lifetest).

5. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy
Description: Time to initiation of cytotoxic chemotherapy was defined as the time from randomization to the date of initiation of cytotoxic chemotherapy for prostate cancer.
Time Frame: Up to approximately 43 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Apalutamide
Number analyzed (Participants) | 401 | 806
Months | NA [NA to NA] — The median was not estimable (NA) as KM curve did not drop to 0.5 or below. The lower or upper limit was NA as lower or upper limit of CI for survivor function was above 0.5 using log(-log) transformation (default of SAS Proc Lifetest). | NA [NA to NA] — The median was not estimable (NA) as KM curve did not drop to 0.5 or below. The lower or upper limit was NA as lower or upper limit of CI for survivor function was above 0.5 using log(-log) transformation (default of SAS Proc Lifetest).

6. Primary Outcome: Metastasis-Free Survival (MFS) by Blinded Independent Central Review (BICR)
Description: MFS was defined as the time from randomization to the time of first evidence of BICR-confirmed bone or soft tissue distant metastasis or death due to any cause, whichever occurred first. The MFS data for participants without metastasis or death were performed for US or ex-US regulatory purposes. Radiographic scans (bone scans and computerized tomography [CT] or magnetic resonance imaging [MRI] of the chest, abdomen, and pelvis) were performed for detection of metastasis throughout the study.
Time Frame: Up to approximately 43 Months
Population: Intent-to-Treat (ITT) population included all participants who were randomized into the study, with study drug assignments designated according to initial randomization, regardless of whether participants received what was assigned.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Apalutamide
Number analyzed (Participants) | 401 | 806
Months
  US Regulatory | 16.20 [14.59 to 18.40] | 40.51 [NA to NA] — NA signifies: lower and upper limit of Confidence Interval(CI) was not estimable as lower, or upper, or both limits of CI for survivor function were above 0.5 using log(-log) transformation (default of Statistical Analysis System[SAS] Proc Lifetest).
  Ex-US Regulatory | 15.70 [14.55 to 18.40] | 40.51 [29.70 to 40.51]
Statistical Analysis 1: Comparison: Placebo vs Apalutamide; Statistical Analysis for MFS by BICR (US Regulatory); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.280, 95% CI 2-sided [0.227 to 0.346]
Statistical Analysis 2: Comparison: Placebo vs Apalutamide; Statistical Analysis for MFS by BICR (Ex-US Regulatory); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.297, 95% CI 2-sided [0.244 to 0.362]

ADVERSE EVENTS:
Time Frame: Up to approximately 43 months
Description: Safety population included all participants who received at least one dose of study drug.
Arm/Group | Placebo | Apalutamide
All-Cause Mortality (participants affected / at risk) | 1/398 | 10/803
Serious Adverse Events (participants affected / at risk) | 92/398 | 199/803
Other Adverse Events (participants affected / at risk) | 329/398 | 716/803
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=398) | Apalutamide (N=803)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Acute Coronary Syndrome (Cardiac disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 1
Angina Unstable (Cardiac disorders) | 0 | 1
Aortic Valve Incompetence (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 7
Atrial Flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 3
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 4
Cardiomyopathy (Cardiac disorders) | 0 | 2
Coronary Artery Disease (Cardiac disorders) | 1 | 3
Coronary Artery Occlusion (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 3
Myocardial Ischaemia (Cardiac disorders) | 1 | 1
Right Ventricular Dysfunction (Cardiac disorders) | 0 | 1
Sinus Node Dysfunction (Cardiac disorders) | 0 | 1
Stress Cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Choroidal Haemorrhage (Eye disorders) | 1 | 0
Open Angle Glaucoma (Eye disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Chronic Gastritis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Enteritis (Gastrointestinal disorders) | 0 | 1
Erosive Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 0 | 1
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal Mass (Gastrointestinal disorders) | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal Achalasia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Dystrophic Calcification (General disorders) | 0 | 1
Gait Disturbance (General disorders) | 1 | 1
General Physical Health Deterioration (General disorders) | 0 | 2
Hyperthermia (General disorders) | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 3
Oedema Peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 5
Soft Tissue Inflammation (General disorders) | 0 | 1
Cholangitis Acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 1
Appendiceal Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 3
Cellulitis Streptococcal (Infections and infestations) | 0 | 1
Cellulitis of Male External Genital Organ (Infections and infestations) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis Clostridial (Infections and infestations) | 0 | 1
H1n1 Influenza (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 2 | 9
Pneumonia Parainfluenzae Viral (Infections and infestations) | 0 | 1
Prostatic Abscess (Infections and infestations) | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 7
Severe Fever with Thrombocytopenia Syndrome (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 0 | 1
Staphylococcal Skin Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 10
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 5
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 | 2
Anastomotic Complication (Injury, poisoning and procedural complications) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Avulsion Fracture (Injury, poisoning and procedural complications) | 1 | 0
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 6
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 3
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 2
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 2
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 2
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 3
Perirenal Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 2
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 2
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 3
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 2
Blood Bilirubin Increased (Investigations) | 0 | 1
Blood Urine Present (Investigations) | 1 | 0
Eastern Cooperative Oncology Group Performance Status Worsened (Investigations) | 0 | 1
Weight Decreased (Investigations) | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 5
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Flattening (Musculoskeletal and connective tissue disorders) | 0 | 1
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Neoplasm of Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant Neoplasm of Renal Pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 2
Balance Disorder (Nervous system disorders) | 0 | 1
Central Nervous System Lesion (Nervous system disorders) | 1 | 0
Cerebellar Infarction (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Lacunar Stroke (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Spinal Cord Compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 5
Thrombotic Cerebral Infarction (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 3
Device Occlusion (Product Issues) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Major Depression (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 4 | 6
Azotaemia (Renal and urinary disorders) | 0 | 1
Bladder Mass (Renal and urinary disorders) | 1 | 0
Bladder Neck Sclerosis (Renal and urinary disorders) | 1 | 0
Bladder Necrosis (Renal and urinary disorders) | 0 | 1
Calculus Urethral (Renal and urinary disorders) | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 1 | 0
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 3
Haematuria (Renal and urinary disorders) | 8 | 13
Hydronephrosis (Renal and urinary disorders) | 8 | 8
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 1 | 0
Micturition Disorder (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 3 | 3
Renal Impairment (Renal and urinary disorders) | 0 | 1
Strangury (Renal and urinary disorders) | 0 | 1
Ureteric Obstruction (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 1
Urethral Stenosis (Renal and urinary disorders) | 1 | 2
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 15 | 10
Urinary Tract Obstruction (Renal and urinary disorders) | 4 | 2
Prostatic Mass (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Granuloma Annulare (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic Aneurysm (Vascular disorders) | 0 | 2
Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypertensive Crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Venous Aneurysm (Vascular disorders) | 0 | 1
Venous Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=398) | Apalutamide (N=803)
Anaemia (Blood and lymphatic system disorders) | 15 | 51
Hypothyroidism (Endocrine disorders) | 5 | 48
Abdominal Discomfort (Gastrointestinal disorders) | 22 | 37
Abdominal Pain (Gastrointestinal disorders) | 33 | 64
Abdominal Pain Upper (Gastrointestinal disorders) | 32 | 44
Constipation (Gastrointestinal disorders) | 52 | 87
Diarrhoea (Gastrointestinal disorders) | 60 | 159
Dyspepsia (Gastrointestinal disorders) | 22 | 58
Nausea (Gastrointestinal disorders) | 63 | 145
Vomiting (Gastrointestinal disorders) | 24 | 43
Asthenia (General disorders) | 33 | 89
Fatigue (General disorders) | 84 | 244
Oedema Peripheral (General disorders) | 29 | 68
Nasopharyngitis (Infections and infestations) | 25 | 78
Upper Respiratory Tract Infection (Infections and infestations) | 21 | 44
Urinary Tract Infection (Infections and infestations) | 37 | 57
Fall (Injury, poisoning and procedural complications) | 35 | 121
Weight Decreased (Investigations) | 25 | 128
Decreased Appetite (Metabolism and nutrition disorders) | 35 | 99
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 49
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 128
Back Pain (Musculoskeletal and connective tissue disorders) | 59 | 100
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 20 | 73
Dizziness (Nervous system disorders) | 25 | 74
Dysgeusia (Nervous system disorders) | 6 | 57
Headache (Nervous system disorders) | 25 | 75
Insomnia (Psychiatric disorders) | 21 | 55
Dysuria (Renal and urinary disorders) | 22 | 41
Haematuria (Renal and urinary disorders) | 34 | 60
Nocturia (Renal and urinary disorders) | 29 | 39
Pollakiuria (Renal and urinary disorders) | 34 | 45
Urinary Incontinence (Renal and urinary disorders) | 15 | 42
Urinary Retention (Renal and urinary disorders) | 24 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 58
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 63
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 50
Rash (Skin and subcutaneous tissue disorders) | 13 | 87
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 | 43
Hot Flush (Vascular disorders) | 34 | 113
Hypertension (Vascular disorders) | 77 | 198

LIMITATIONS AND CAVEATS:
These results are up to clinical cutoff (CCO) date (that is, 19 May 2017).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT01946204/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT01946204/SAP_001.pdf